CLINICAL TRIAL: NCT00568061
Title: The Effects of Nitric Oxide for Inhalation on Myocardial Infarction Size
Brief Title: Nitric Oxide in Myocardial Infarction Size
Acronym: NOMI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INOT 44
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2010-08-27 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2016-05

CONDITIONS: Acute Myocardial Infarction; ST Elevation MI; STEMI
Keywords: INOT44; NOMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): Inhaled Nitric oxide administered at 80 parts per million (ppm)
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Inhaled nitrogen gas (Placebo) administered at 80 ppm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Nitric oxide for inhalation
  Other Names: INOmax®
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Nitrogen gas (placebo) for inhalation
  Other Names: Nitrogen gas
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether or not inhaled nitric oxide can decrease myocardial infarction (MI) size at 48-72 hours in patients presenting with an ST segment elevation MI (STEMI) who undergo successful percutaneous coronary intervention.

DETAILED DESCRIPTION:
The purpose of the trial is to assess whether or not inhaled nitric oxide can decrease myocardial infarction (MI) size as a fraction of left ventricular (LV) size at 48-72 hours in patients presenting with an ST segment elevation MI who undergo successful percutaneous coronary intervention (PCI).

The primary endpoint for this study will be myocardial infarction size as a fraction of left ventricular size at 48-72 hours as measured by contrast-enhanced cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction and electrocardiographic evidence of ST elevation
* No clinical evidence of congestive heart failure
* All patients must undergo successful percutaneous coronary intervention for thrombolysis in myocardial infarction (TIMI) 0 or 1 coronary flow with resulting TIMI 2 or 3 flow
* Greater than 18 years of age
* Signed Institutional Review Board (IRB) approved informed consent

Exclusion Criteria:

* Prior myocardial infarction
* Requirement for urgent cardiac surgery
* Previous coronary artery bypass graft (CABG) or primary coronary intervention (PCI)
* Left bundle branch block
* Heart block that is expected to require a temporary pacemaker for greater than 72 hours
* Prior use of thrombolytic therapy for the current event
* Unable to tolerate magnetic resonance imaging or unable to tolerate gadolinium contrast media, including patients with a calculated creatinine clearance less than 60 ml/min/1.73m² Body Surface Area (BSA)
* Active or recent hemorrhage requiring an invasive procedure for evaluation or transfusion within 6 weeks prior to presentation, or hemorrhagic stroke within the 6 weeks prior
* Neutropenia (WBC <2000 (mm)³), Anemia (HCT <30%, Thrombocytopenia (Thrombocytes <50,000 (mm)³). It is not necessary to confirm blood counts prior to start of study drug in the absence of clinical suspicion.
* Known or suspected aortic dissection.
* Prior history of pulmonary disease requiring chronic oxygen therapy.
* Pregnancy, lactating, and women of childbearing potential.
* Medical problem likely to preclude completion of the study.
* Use of investigational drugs or device within the 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Baldassarre, MD, Study Director — Mallinckrodt
Locations (14):
- United States (11):
  - Providence Hospital, Mobile, Alabama
  - Baptist Cardiac & Vascula Institute, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jack D. Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - LeBauer Cardiology, Greensboro, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Central Utah Imaging, Provo, Utah
- Virga Jesse Hospital, Hasselt, Belgium
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 medical centers enrolled subjects. A total of 29 subjects were enrolled in the study.
Groups:
- Inhaled Nitric Oxide: Inhaled Nitric Oxide administered at 80 ppm
- Nitrogen Gas: Nitrogen Gas (Placebo) administered at 80 ppm
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Started | 13 | 16
Completed | 8 | 14
Not Completed | 5 | 2
Not completed — Inclusion / exclusion criteria | 5 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide: Inhaled Nitric Oxide administered at 80ppm
- Nitrogen Gas: Nitrogen Gas (Placebo) administered at 80ppm
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.71) | 63.8 (12.41) | 63.1 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Myocardial Infarction Size to the Fraction of Left Ventricular Size
Description: The primary endpoint - mean percent of the myocardial infarction size to the fraction of left ventricular size at 48-72 hours was measured by contrast-enhanced cardiac Magnetic Resonance Imaging (MRI).
Time Frame: 48-72 hours
Population: Analysis was per intent to treat population
Measure: Mean (Standard Deviation); unit: percent of myocardial infarction size
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 13 | 16
percent of myocardial infarction size | 15.8 (8.99) | 12.5 (11.68)

2. Secondary Outcome: Myocardial Infarction (MI) Size at 48-72 Hours
Time Frame: 48-72 hours
Population: All efforts have been exhausted to locate data for this historical trial - the validated summary tables and Clinical Study Report (CSR) are no longer accessible.
Arm/Group | Nitric Oxide
Number analyzed (Participants) | 0

3. Secondary Outcome: MI Size Normalized to Area at Risk
Time Frame: 48-72 hours
Population: All efforts have been exhausted to locate data for this historical trial - the validated summary tables and CSR are no longer accessible.
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Myocardial Perfusion at Coronary Angiography
Time Frame: at completion of primary coronary intervention (PCI)
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Infarct Transmurality
Time Frame: 48-72 hours and 4 months
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Global & Regional Left Ventricular (LV) Function and LV Mass
Time Frame: 48-72 hours and 4 months
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Global LV Function and Mass
Time Frame: between 48-72 hours and 4 months
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: MI Size as a Fraction of LV Size
Time Frame: 4 months
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Resolution of ST Segment Elevation Compared With That Observed at Enrollment
Time Frame: 4 hours
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Troponin T Levels and CPK-MB Area Under the Curve
Time Frame: 48 hours
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Adverse Remodeling Parameters Compared With 48-72 Hrs: Changes in LV End-diastolic Vol, End-systolic Vol, End-diastolic Myocardial Wall Thickness in Infarct, Peri-infarct and Remote Areas, and in Sphericity Index at End-diastole and End-systole
Time Frame: 4 months
Population: as for outcome 3
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Inhaled Nitric Oxide | Nitrogen Gas
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/16
Other Adverse Events (participants affected / at risk) | 2/13 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=13) | Nitrogen Gas (N=16)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Retropertioneal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=13) | Nitrogen Gas (N=16)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The validated summary tables and CSR are not available for this legacy registration that was transferred to us eight years after it was terminated for low enrollment, so posting of results for secondary outcome measures is not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No